CLINICAL TRIAL: NCT00722501
Title: Ascending Single Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ERB-257 Administered Intravenously as a 30-Minute Infusion to Healthy Subjects
Brief Title: Study Evaluating the Safety and Pharmacokinetics of Ascending Single IV Doses of ERB-257
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3252K1-1000
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2009-04-28 (Estimated); Status verified 2009-04

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ERB-257 (Active Comparator): 7 IV single doses of ERB-257 will be given to 6 healthy subjects per group - 1,4, 15, 45, 90, 180, and 300 mg
  Interventions: Drug: ERB-257
- placebo (Placebo Comparator): 2 placebo subjects per group
  Interventions: Other: placebo

INTERVENTIONS:
Drug: ERB-257
  Arms: ERB-257
Other: placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of ascending single IV doses of ERB-257 in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women of non-childbearing potential between the ages of 18 and 50.
2. Body mass index (BMI) in the range of 18.0 to 30.0 kg/m2 and body weight greater than or equal to 50 kg2.
3. Have a high probability for compliance with and completion of the study.

Exclusion Criteria:

1. Presence or history of any disorder that may prevent the successful completion of the study.
2. Acute disease state (eg, nausea, vomiting, fever, or diarrhea) within 7 days before study day 1.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2008-08; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of single ascending IV doses of ERB-257 administered to healthy subjects | 4 days per group

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics of single ascending IV doses of ERB-257 administered to healthy subjects | 4 days per group

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Trial Manager, Philadelphia, Pennsylvania, United States